CLINICAL TRIAL: NCT05617586
Title: Early Development and Diagnostic Trajectories in the Child With DCD in Flanders
Brief Title: Early Development and Diagnostic Trajectories in DCD
Acronym: DCD_Parent
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201836914
Record Dates: First submitted 2019-01-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Developmental Coordination Disorder
Keywords: Early Development; Diagnostic trajectory; Parental report; Qualitative study
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCD Parents: An in-depth interview will be conducted of parents of a child with DCD. Parents will be asked to complete a Developmental Coordination Disorder Questionnaire (DCD-Q).
  Interventions: Other: In-depth parental interview; Other: Developmental Coordination Disorder Questionnaire (DCD-Q)

INTERVENTIONS:
Other: In-depth parental interview — A semi-structurerd interview will be conducted of parents with a child diagnosed with DCD. The interview will be audio-recorderded. The audiofile will be transcribed ad-verbatim and analyzed using narrative analysis methods.
Other: Developmental Coordination Disorder Questionnaire (DCD-Q) — Parents will be asked to complete the DCD-Q. This will help us describe the sample.

SUMMARY:
The aim of this study is to map the early development of children with DCD and the diagnostic trajectory in Flanders.

DETAILED DESCRIPTION:
The Diagnostic and Statistical manual 5th edition (DSM-V) defines Developmental Coordination Disorder (DCD) as early-onset deficits in acquiring and executing motor coordination skills. These deficits significantly interfere with the performance of activities of daily living and impact on academic productivity, leisure and play.

Although DCD can be identified during preschool, diagnosis generally occurs at primary-school age. Before the age of three (t.i. infancy), some parents already express "something is wrong" with their child albeit DCD is rarely diagnosed within this age-group.

Knowledge on DCD in children before the age of five is limited. The aim of this study is twofold: to explore the early development of children with DCD and to map the diagnostic trajectory of DCD in Flanders.

Design: A qualitative narrative inductive study design by means of audio-recorded in-depth interviews

Sampling: Purposeful maximum variation sampling will be applied.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or guardian of a child diagnosed with DCD
2. Diagnosis of DCD within the last two years
3. Child was max. 12y of age at the moment of DCD diagnosis

Exclusion Criteria:

1. No severe diseases in early childhood greatly impacting development (cancer, severe accident,…)
2. Diagnosis outside of Belgium

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children with DCD
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Early Developmental characteristics of children with DCD during pregnancy (qualitative research) by means of an interview. | 20 interviews (duration: approximately 1.5 to 2 hours) starting from january 2019 to december 2020
  As we will conduct a qualitative narrative analysis of the interviews, no standardised measurement tools will be used.
  We will probe for the following fields of interest:
  - Pregnancy:(fetal movements, birth complications)
Early Developmental characteristics of children with DCD during toddlerhood (qualitative research) by means of an interview. | 20 interviews (duration: approximately 1.5 to 2 hours) starting from january 2019 to december 2020
  As we will conduct a qualitative narrative analysis of the interviews, no standardised measurement tools will be used.
  We will probe for the following fields of interest:
  - Todderhood (feeding, cyring, sleeping, milestones, behavior, play)
Early Developmental characteristics of children with DCD (preschooler) (qualitative research) by means of an interview. | 20 interviews (duration: approximately 1.5 to 2 hours) starting from january 2019 to december 2020
  As we will conduct a qualitative narrative analysis of the interviews, no standardised measurement tools will be used.
  We will probe for the following fields of interest:
  - Preschooler (interests, motor activities, behavior, friends, fatigue, communication, play)

SECONDARY OUTCOMES:
Diagnostic trajectories of children with DCD in Flanders by means of an interview. | 20 interviews (duration: approximately 1.5 to 2 hours) starting from january 2019 to december 2020
  As we will conduct a qualitative narrative analysis of the interviews, no standardised measurement tools will be used.
  We will probe for the following field of interest:
  * Did parents/creche/family/friends/school express concerns which have led to seeking advice/help? Which concerns?
  * Which advises or what help did parents receive from who? What did they do with them?
  * Which caregivers did they consult? What were the results/advices?
  * Who diagnosed the child with DCD? Who was involved?
  * Which elements led to the diagnosis of DCD?
  We will map the trajectories leading to a diagnosis of DCD in Flanders.

CONTACTS AND LOCATIONS:
Overall Officials: Amy De Roubaix, Master, Principal Investigator — University Ghent; Hilde Van Waelvelde, PhD, Study Chair — University Ghent; Dominique Van De Velde, PhD, Study Chair — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No